CLINICAL TRIAL: NCT02621918
Title: The Effects of an Intradialytic Progressive Resistance and Aerobic Training in End-stage Renal Disease Patients Undergoing Hemodialysis
Brief Title: The Effects of Exercise in End-stage Renal Disease Patients Undergoing Hemodialysis
Acronym: EESRDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Clara S C Rosa, PhD Student, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CAAE-02564112.2.0000.5423
Record Dates: First submitted 2015-10-21; First posted 2015-12-04 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Renal Failure on Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Progressive Resistance Training (PRT) (Experimental): For the progressive resistance training we use 11 exercises. The exercises for upper limbs were held in the waiting room before the hemodialysis session. Resistance exercise was carried out in two sets of 15-20 repetitions, the intensity were determined by the method of maximal repetitions, where series were run until exhaustion to momentary exercises (15-20 repetitions) with specific load. The load adjustments or volume were managed when necessary, but necessarily for every 4th week of training. The effort perception should be situated between 12 and 16 on the Borg scale (Borg and Noble, 1974), as proposed by The Life Options Rehabilitation Advisory Council: Exercise for the Patient Dialysis (1995).
  Interventions: Other: Progressive resistance training
- Aerobic Exercise (AER) (Experimental): Aerobic exercise was conducted with a mini ergometer cycling (Mini Bike E5 Acte Sports) attached to the patient chair. Patients exercised 50-60 minutes of continuous workout with increased load. The workload was adjusted when necessary, according to the perceived effort made by the patient. The scale of perceived exertion, Borg scale (Borg and Noble , 1974), was used in accordance with the proposed By The Life Options Rehabilitation Advisory Council: Exercise for the Patient Dialysis (1995), which defines the values of perceived exertion between 12 and 16.
  Interventions: Other: Aerobic training
- NEPLA (Placebo Comparator): The control group performed active mobilization of members, circumduction of cervical, scapular girdle and extremities, breathing exercises with no loads, set on three to five repetitions only and no stretch exercises. The exercises were performed during the hemodialysis session, three times per week and did not exceed 5 minutes.
  Interventions: Other: Placebo training

INTERVENTIONS:
Other: Progressive resistance training
  Arms: Progressive Resistance Training (PRT)
Other: Aerobic training
  Arms: Aerobic Exercise (AER)
Other: Placebo training
  Arms: NEPLA

SUMMARY:
We aimed to investigate the effect of a progressive resistance training and aerobic training protocol on functional capacity, body composition and quality of life.

DETAILED DESCRIPTION:
Subjects were randomized into group A and B: group A (n=30) exercised for the first 6 months while group B (n=31) performed a placebo exercise initially (3 months) and cross-over to aerobic exercised for 3 months more.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years
* more than three months of hemodialysis vintage
* under the permission of their nephrologist
* agreement to be randomly assigned and undergo study protocols

Exclusion Criteria:

* Patients in wheelchair, presenting disability, or those who had amputation and malformation of the lower limbs, causing impaired walking
* presenting representative blindness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-03; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Body composition by Dual-energy x-ray absorptiometry (DEXA) | before and after 12 and 24 weeks of study
  Dual-energy x-ray absorptiometry (DEXA) was used to measure lean body mass (LBM), fat mass (FM) and Bone Mineral Contend (BMC) in grams using a total body scan, following the equipment description - HOLOGIC Discovery Wi (Hologic inc, Waltham, MA, USA). Body composition variables included in this study were total mass, body FM, LBM and legs LBM, and BMC. Body composition was assessed after a hemodialysis day; time after previous hemodialysis did not exceed eight hours.

SECONDARY OUTCOMES:
Quality of life assessed by the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36) | before and after 12 and 24 weeks of study
  Quality of life assessment was analyzed using the Medical Outcomes Study 36-item Short-Form Health Survey (SF-36). The SF-36 is composed of eleven issues of 36 items that assess eight dimensions events occurred in the last four weeks. For the presentation of the survey results, the final score of each domain was transformed into a scale from 0 (worse) to 100 (better). Total score, mental e physical dimensions were analyzed separated.
Functional capacity | before and after 12 and 24 weeks of study
  The 6 minutes walking test measured the walking capacity (distance in meters) during 6 minutes. The sit-to-stand test assessed the lower limbs strength resistance by times that the subject stand and sit (chair) during 30 seconds. And flexibility was assessed by sit and reach test.
Pulmonary capacity | before and after 12 and 24 weeks of study. Additionally this variable was assessed over the three time points before and after one hemodialysis session.
  For the assessment of maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) an analog manovacuometer (Gerar ®, 0±300 cmH2O) was used. Patients underwent three valid maneuvers and the most negative and most positive in MIP and MEP, respectively, were considered. Ventilometer (Ferraris Mark8 Wright Respirometer®) detected the low vital capacity (LVC). Reduced forced expiratory volume in one second (FEV1), reduced forced vital capacity (FVC), normal FEV1/FVC ratio, and forced expiratory flow between 25% and 75% of vital capacity (FEF25-27) were evaluated with the spirometer brand IQTeQ. Spirometric variables were analyzed in reference percentage values in order to eliminate the effects of age, height, and gender. The assay was performed in order to obtain three acceptable curves with at least two reproducible curves five minutes interval for each exam for a total of up to eight trials.

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639